CLINICAL TRIAL: NCT03688113
Title: The Use of a Smartphone Application for Tinnitus Treatment
Brief Title: Tinnitus Treatment Using a Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Director, Research and Development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0493-18-TLV
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Tinnitus application
- Wait list (Other)
  Interventions: Behavioral: Tinnitus application

INTERVENTIONS:
Behavioral: Tinnitus application — Use of tinnitus application

SUMMARY:
People with tinnitus will use a smartpphone app in which they are instructed to reject maladaptive thoughts by throwing them away from themselves (upwards) and embrace supportive thoughts by pulling them towards themselves (downwards). The Tinnitus Handicap Inventory will be used to measure the effect of the application.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus lasting more than 3 months

Exclusion Criteria:

* Brain space occupying lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory score | 34 days
  The Tinnitus Handicap Inventory measures the degree of disturbance the tinnitus causes the patients, on a a total scale of 0-100. 0 is the lowest possible score (no disturbance caused by the tinnitus, 100- the most severe form of intrusiveness)

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No